CLINICAL TRIAL: NCT01512381
Title: Variant of Stimulation in Atrioventricular Node Ablation (VISTA) in Patients With Atrial Fibrillation and Moderate Chronic Heart Failure
Brief Title: Atrioventricular Node Ablation in Patients With Atrial Fibrillation and Moderate Chronic Heart Failure
Acronym: VISTA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Absence of patients for recruitment
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: zubarev-vista-17-12
Record Dates: First submitted 2012-01-12; First posted 2012-01-19 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2017-01

CONDITIONS: Heart Failure
Keywords: heart failure; CRT; atrial fibrillation; AV junction ablation
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CRT (Experimental)
  Interventions: Device: Implantation of CRT device
- pacemaker (Active Comparator)
  Interventions: Device: Implantation of conventional VVI(R) pacemaker

INTERVENTIONS:
Device: Implantation of CRT device — RV lead of CRT system is implanted into the middle part of interventricular septum
  Arms: CRT
Device: Implantation of conventional VVI(R) pacemaker — RV lead is implanted into the middle part of interventricular septum
  Arms: pacemaker

SUMMARY:
The purpose of this study is to determine whether cardiac resynchronization therapy (CRT) is superior to interventricular right ventricle (RV) septal pacing in respect of reverse remodeling (LV ESD) and morbidity in patients with less preserved (less than 45%) ejection fraction (EF), persistent/permanent atrial fibrillation (AF) who successfully received atrioventricular (AV) junction ablation ablation (100% pacemaker dependency)

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-75 years
* CHF II-III NYHA
* Persistent/permanent AF requiring AV node ablation
* LVEF < 45%
* Signed informed consent
* Able to complete all testing required by the clinical protocol

Exclusion Criteria:

* Myocardial infarction or stroke less than 3 months prior to randomization
* Patients who require revascularization, radiofrequency ablation of pulmonary veins and substrate of AF
* The congenital and acquired heart diseases, LV aneurysm, which requires a surgical correction
* Active inflammatory and autoimmune diseases of a myocardium
* The thyrotoxicosis
* The diseases that limit life expectancy (cancer, tuberculosis, etc.)
* Contraindications to anticoagulants administration at CHADS2> 2
* Uncompliant patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Left Ventricle End-Systolic Volume (LV ESV) | 12 months

SECONDARY OUTCOMES:
Rate of cardiovascular events (hospitalization for worsening heart failure) | 12 month
Changes in Quality of Life (measured by Minnesota Living with Heart Failure Questionnaire) | 12 months
Changes in NYHA functional class measured by peak V O2 oxygen consumption and distance of 6-minute walk test | 12 months
Echocardiographic indexes of LV remodeling | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Almazov Federal Heart, Blood and Endocrinology Centre, Saint Petersburg, Russia